CLINICAL TRIAL: NCT01733810
Title: The Role of HIF-2a in the Pathogenesis of Reflux Esophagitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Stuart Spechler, Professor of Medicine, Dallas VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2R01DK063621-11 (NIH); R01DK063621 (NIH)
Record Dates: First submitted 2012-11-16; First posted 2012-11-27 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Esophagitis; Reflux Esophagitis; Gastroesophageal Reflux Disease
Keywords: Esophagitis; Reflux esophagitis; Gastroesophageal reflux disease; Acid; Inflammation; Esophagus; Cytokines; Esophageal squamous cell; Reflux; Squamous epithelium
MeSH Terms: conditions — Esophagitis; Esophagitis, Peptic; Gastroesophageal Reflux; Heartburn; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reflux Patients (Experimental): Patients with reflux and a prior history of reflux esophagitis are being enrolled. The intervention is cessation of acid-suppressing medications.
  Interventions: Other: Cessation of Acid Suppressing Medications

INTERVENTIONS:
Other: Cessation of Acid Suppressing Medications — Acid-suppressing medications are stopped for all participants the day after baseline assessment. Subsequent evaluations performed while participant is not on acid-suppressing medications.

SUMMARY:
The purpose of this study is to determine the role of hypoxia inducible factor (HIF)-2a on the production of inflammatory cytokines that lead to reflux esophagitis.

DETAILED DESCRIPTION:
Reflux esophagitis is thought to be caused by gastric acid that refluxes into the esophagus, causing injury. Newer data suggest that reflux of gastric juice into the esophagus stimulates HIF-2a, which increases production of inflammatory cytokines. These cytokines are thought to lead to reflux esophagitis. The investigators plan to study the relationship of HIF-2a to inflammatory cytokines in patients with known gastroesophageal reflux disease and reflux esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* U.S Veteran
* History of Los Angeles Grade C erosive esophagitis

Exclusion Criteria:

* Inability to provide informed consent
* Esophageal varices
* Warfarin use
* Coagulopathy that precludes safe biopsy of the esophagus
* Comorbidity that precludes safe participation in the study
* Allergy to fluorescein sodium
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
change in esophageal inflammation from baseline to 14 days | day 0 and day 14
  inflammation of the squamous esophageal mucosa will be measured at baseline and at 14 days

SECONDARY OUTCOMES:
change in HIF-2a levels from baseline to 14 days | day 0 and day 14
  Amount of HIF-2a present will be measured at baseline and at 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Spechler, MD, Principal Investigator — Dallas VA Medical Center
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Huo X, Agoston AT, Dunbar KB, Cipher DJ, Zhang X, Yu C, Cheng E, Zhang Q, Pham TH, Tambar UK, Bruick RK, Wang DH, Odze RD, Spechler SJ, Souza RF. Hypoxia-inducible factor-2alpha plays a role in mediating oesophagitis in GORD. Gut. 2017 Sep;66(9):1542-1554. doi: 10.1136/gutjnl-2016-312595. Epub 2016 Sep 30. PMID 27694141
- [Derived] Dunbar KB, Agoston AT, Odze RD, Huo X, Pham TH, Cipher DJ, Castell DO, Genta RM, Souza RF, Spechler SJ. Association of Acute Gastroesophageal Reflux Disease With Esophageal Histologic Changes. JAMA. 2016 May 17;315(19):2104-12. doi: 10.1001/jama.2016.5657. PMID 27187303